CLINICAL TRIAL: NCT03318263
Title: Monitoring of ESR1, PIK3CA and AKT ctDNA Mutations During Real-life Followup of Patients With Metastatic Breast Cancer Treated With Aromatase Inhibitors
Brief Title: CIrCuLAting Dna ESr1 Gene Mutations Analysis
Acronym: CICLADES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A01767-46
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: Estrogen-receptor-positive breast cancer; aromatase inhibitor,; ESR1,; PIK3CA; AKT; endocrine resistance; circulating tumor DNA
MeSH Terms: conditions — Breast Neoplasms; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Other)
  Interventions: Diagnostic Test: next-generation sequencing (NGS)

INTERVENTIONS:
Diagnostic Test: next-generation sequencing (NGS) — ESR1, PI3KCA and AKT extensive exon sequencing will be performed using NGS (Miseq Illumina) at the Biopathology department, Institut de Cancérologie de Lorraine (ISO15189 certified lab). Samples taken at baseline (t0), at progression (tp) and 3 months before progression (tp-3) will be systematically analyzed. The intermediate samples will be stored and kept for additional studies. Follow up assessment will be performed according to prescriber's directions.

SUMMARY:
The estrogen-dependent nature of breast cancer was first reported in 1896 with the publication of George Beatson's observations on the regression of breast cancer following oophorectomy. Endocrine therapy, targeting ER either directly by selective estrogen receptor modulators (SERMs) and pure antagonists or indirectly by aromatase inhibitors (AIs) that block estrogen production, remains the mainstay of treatment of hormone-sensitive breast cancer in the adjuvant and metastatic settings.

Intrinsic (de novo) and acquired endocrine resistance constitutes an important clinical challenge in the treatment of breast cancer and multiple mechanisms are suspected to underlie the emergence of endocrine resistance.

The role of the estrogen receptor (ER), encoded by the ESR1 gene, in normal mammary gland development and the progression of breast cancer is well established. ESR1 mutations, occurring in 10 to 30% of ER-positive metastatic breast cancer resistant to AIs, lead to ligand-independent activation of the ER.

For patients treated with AIs, monitoring of circulating tumour DNA (ctDNA) for ESR1, PIK3CA and AKT1 mutations could permit early detection of resistance to AIs as recently reported during 2016 American Society of Clinical Oncology (ASCO) meeting.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient aged 18 and older
2. Histologically confirmed estrogen-receptor-positive, HER2-negative breast cancer
3. Proven metastatic (AJCC stage IV) or loco-regionally advanced (AJCC stage III) breast cancer, not amenable to surgery or radiation with curative intent.
4. Indication to treat with first-line endocrine therapy for palliative care.

   * Patients already receiving first-line endocrine therapy can be enrolled up to 6 weeks after start of endocrine therapy.
   * Endocrine therapy can be prescribed in combination with a CDK4/6 inhibitor.
   * One prior regimen of chemotherapy for the treatment of advanced disease is allowed.
   * Prior (neo)adjuvant chemotherapy and/or (neo)adjuvant endocrine therapy is/are allowed; patients with recurrence while on adjuvant endocrine therapy can be enrolled.
5. Patients who can benefit from an additional blood sample of 10ml. The total volume of each sample meets with the indications of the Order in force establishing the list of researches mentioned in 2 ° of Article L. 1121-1 of the Public Health Code.
6. Informed consent explained to, understood by and signed by patient. Patient must be given a copy of informed consent.
7. Patients affiliated to a social security scheme or benefit from a social regime

The prescription of medicinal product(s) is clearly separated from the decision to include the subject in this ISMRC.

Exclusion Criteria:

1. Pregnant or breast-feeding woman.
2. Patient who received any prior systemic hormonal therapy for advanced breast cancer; no more than one prior regimen of chemotherapy for the treatment of advanced disease is allowed.
3. Chemotherapy in combination with endocrine therapy.
4. Targeted therapy, except CDK 4/6 inhibitor, in combination with endocrine therapy.
5. Planned surgery or radiation with curative intent.
6. Other active malignancy.
7. Any concurrent severe and/or uncontrolled medical condition(s) which could compromise participation in the study.
8. Patient whose general state and / or conditions do not permit the collection of the additional blood sample.
9. Patients under guardianship, under curatorship or deprived of liberty.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
incidence of ESR1 mutations | 1 day

SECONDARY OUTCOMES:
incidence of PIK3CA and AKT1 mutations | 1 day
prevalence of ESR1, PIK3CA and AKT1 mutations in patients with and without endocrine resistance at enrolment | 1 day
prevalence of ESR1, PIK3CA and AKT1 mutations in patients according to mono vs combo therapy. | 1 day
prevalence of mutations of other genes of interest included in the panel from the start of treatment to progression or end of follow-up | 1 day
ESR1, PIK3CA and AKT1 mutations predictor of progression free survival | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: MASSARD VINCENT, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (10):
- France (10):
  - Hôpital Claude Bernard, Metz
  - CHR Metz-Thionville, Metz
  - Centre d'oncologie Gentilly, Nancy
  - Institut Jean Godinot, Reims
  - Polyclinique de Courlancy, Reims
  - Centre Henri Becquerel, Rouen
  - Polyclinique de l'Orangerie, Strasbourg
  - Clinique Saint Anne, Strasbourg
  - CHU Strasbourg, Strasbourg
  - Institut de cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No